CLINICAL TRIAL: NCT07174284
Title: CAN TRUNK IMPAIRMENT LEVEL AND UPPER EXTREMITY FUNCTIONAL CAPACITY IN STROKE SURVIVORS IN THE ACUTE PERIOD PREDICT TRUNK RECOVERY IN THE SUBACUTE PERIOD?
Brief Title: Trunk Impairment and Upper Extremity Function
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Emre Şenocak, Asisstant Professor, Karadeniz Technical University
Other Study IDs: 2024/76
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Prediction; Upper Extremity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Strokers: Individuals with early-stage stroke were included in the study.
  Interventions: Other: No Intervention: Observational Cohort

INTERVENTIONS:
Other: No Intervention: Observational Cohort — No intervention was applied to the patients within the scope of this study.

SUMMARY:
This study examines whether early-term upper extremity functions of acute stroke patients can be a tool for predicting later-period trunk functions.

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 30-80 years with a confirmed diagnosis of ischemic or hemorrhagic stroke were considered for participation.

Exclusion Criteria:

- Patients with secondary orthopedic and/or neurological conditions, lumbosacral injuries, impaired consciousness, unilateral neglect, recurrent stroke, or a Mini-Mental State Examination score <24 were excluded from the study.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute Strokers
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Trunk Impairment Scale | Baseline
  Three items of the scale assess static sitting balance, ten assess dynamic sitting balance, and four assess trunk coordination. The maximum score that can be obtained from these three sections is 23 points.
Trunk Impairment Scale | 30 days after Baseilne assessment
  Three items of the scale assess static sitting balance, ten assess dynamic sitting balance, and four assess trunk coordination. The maximum score that can be obtained from these three sections is 23 points.
Wolf Motor Function Test | Baseline
  The test is a performance tool consisting of seventeen items designed to evaluate the motor skills of the upper extremity. While fifteen items assess functional skills, two items determine muscle strength. Muscle strength was not used in this study. A total score was calculated for the patients' functional skills. The test is scored between 0-5, and the total score varies between 0-75 points for this study

CONTACTS AND LOCATIONS:
Locations (1):
- Bağcılar Training and Research Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided